CLINICAL TRIAL: NCT00545467
Title: Evaluation of the Strategies of Switching Schizophrenia Patients to Aripiprazole From Other Antipsychotic Agents: Combination of Pharmacogenomics and Therapeutic Drug Monitoring
Brief Title: Evaluation of the Strategies of Switching Schizophrenia Patients to Aripiprazole From Other Antipsychotic Agents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Taoyuan Psychiatric Center, Ministry of Health and Welfare, Executive Yuan, R.O.C. Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200705030M
Record Dates: First submitted 2007-10-15; First posted 2007-10-17 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-01

CONDITIONS: DSM-IV Schizophrenia; Schizoaffective Disorder
Keywords: Aripiprazole; schizophrenia; antipsychotics; pharmacogenomics; cytochrome P450 enzyme
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): fast tapering of the previous medication within 1 week after initiating aripiprazole for 2 weeks
  Interventions: Drug: Aripiprazole
- 2 (Active Comparator): slow tapering of the previous medication within 4 weeks after initiating aripiprazole for 2 weeks
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole will be given as a fixed does, 15 mg/day, orally throughout 8 weeks in the 2 arms.
  Other Names: abilify

SUMMARY:
The purpose of this study is to determine whether moderately ill Asian schizophrenic patients can be switched from their previous antipsychotic medication to aripiprazole with minimal adverse clinical consequences, and elucidate both pharmacokinetic and pharmacodynamic factors associated with clinical efficacy of aripiprazole.

DETAILED DESCRIPTION:
Aripiprazole (commercial name abilify) is the first commercially available drug with dopamine partial agonist effects approved for the treatment of schizophrenia and bipolar disorder since 2002 in the U.S. It reduces negative symptoms of schizophrenia efficiently and has a markedly lower incidence of extrapyramidal symptoms and tardive dyskinesia. However, the process of switching other antipsychotic agents to aripiprazole can result in a re-emergence or worsening of psychosis, along with unpleasant side effects such as insomnia, nausea, vomiting, anxiety and agitation. On the basis of a prior study demonstrating the efficacy and safety of aripiprazole in Taiwan population, we hence propose to apply a combined use of pharmacogenomics and therapeutic drug monitoring in the evaluation of the strategies of switching stable schizophrenia patients to aripiprazole from other antipsychotic agents.

We will evaluate their cytochrome P450 background along with other potential candidate genes of schizophrenia. This 2-year proposal will examine the relative efficacy, safety and tolerability of two different strategies for switching stable inpatients/outpatients from prior antipsychotic monotherapy to aripiprazole 15 mg/day monotherapy using two different strategies:

1. Fast tapering of the previous medication within 1 week after initiating aripiprazole for 2 weeks.
2. Slow tapering of the previous medication within 4 weeks after initiating aripiprazole for 2 weeks.

A total of 200 stable schizophrenia patients will be randomized with open label to two strategies.

We expect to achieve the following results:

1. Developing a protocol that has high probability of switching successfully schizophrenia patients to aripiprazole, which is effective in treatment refractory cases and has a markedly lower incidence of severe side effects, from other antipsychotics.
2. Elucidate both pharmacokinetic and pharmacodynamic factors associated with clinical efficacy of aripiprazole.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-lactating, non-pregnant women who are aged 18 to 65 years
* primary diagnosis of DSM-IV schizophrenia or schizoaffective disorder
* taking a stabilized dose of a single oral antipsychotic for at least 1 month prior to study entry
* cannot have been hospitalized for an exacerbation of schizophrenia or schizoaffective disorder for at least 2 months

Exclusion Criteria:

* having other psychiatric disorders
* hospitalizing for acute exacerbation of patients' condition within 2 months
* having taken a selective serotonin reuptake inhibitor (SSRI) within 4 weeks of screening
* a first episode of schizophrenia or schizoaffective disorder
* a clinically significant neurological abnormality other than tardive dyskinesia or EPS
* current diagnosis of psychoactive substance dependence or a historical drug or alcohol abuse within 1 month before the beginning of the study
* treatment with an investigational drug within 4 weeks prior to randomization
* requiring to take medication that inhibits the microsomal enzyme CYP2D6 or inhibits or acts as a substrate for CYP3A4

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-08; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy was assessed using PNASS, Clinical Global Impression (CGI) Scale, and EPS rating scales | on days 0, 7, 14, 28, 56

SECONDARY OUTCOMES:
HPLC analysis Genotyping | on days 0, 14, 56

CONTACTS AND LOCATIONS:
Overall Officials: Tzung-Jeng Hwang, MD, Study Chair — Department of Psychiatry, National Taiwan University Hospital
Locations (1):
- Department of Psychiatry, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Ma CH, Chan HY, Hsieh MH, Liu CC, Liu CM, Hwu HG, Kuo CH, Chen WJ, Hwang TJ. Identifying dopamine supersensitivity through a randomized controlled study of switching to aripiprazole from other antipsychotic agents in patients with schizophrenia. Ther Adv Psychopharmacol. 2022 Jan 28;12:20451253211064396. doi: 10.1177/20451253211064396. eCollection 2022. PMID 35111295
- [Derived] Jen YW, Hwang TJ, Chan HY, Hsieh MH, Liu CC, Liu CM, Hwu HG, Kuo CH, Lin YT, Chien YL, Chen WJ. Abnormally low prolactin levels in schizophrenia patients after switching to aripiprazole in a randomized trial: a biomarker for rebound in psychotic symptoms? BMC Psychiatry. 2020 Nov 23;20(1):552. doi: 10.1186/s12888-020-02957-7. PMID 33228575